CLINICAL TRIAL: NCT02713607
Title: Lipidome and Microbiome Profile of Acne
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 867744
Record Dates: First submitted 2016-03-02; First posted 2016-03-21 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- doxycycline (Experimental): Given doxycycline and assessment of gut, blood and skin
  Interventions: Drug: Doxycycline
- Control (No Intervention): Control subjects to assess if there is baseline difference in these micro-evironments.

INTERVENTIONS:
Drug: Doxycycline — Given doxycycline to acne subjects
  Arms: doxycycline

SUMMARY:
Lipidome and microbiome analysis in subjects with acne on doxycycline. Investigators will look at the skin lipidome, blood lipidome, gut micro biome and skin micro biome.

Investigators will look at the changes between acne subjects and control participants, but also the changes that occur after the use of antibiotics and how this is altered.

DETAILED DESCRIPTION:
We will look at acne subjects, and controls.

We will look at four things

1. skin lipidome
2. skin microbiome
3. gut microbiome
4. blood lipidome

Investigators will assess this in acne participants before and after doxycycline and compare them to controls.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 and older
* Subjects/parents/legal guardian is able to read and comprehend study procedure and consent forms.
* Have already been prescribed Doxycycline by their physician for acne or to be eligible to be prescribed Doxycycline for acne
* Have acne that is diagnosed by a board certified dermatologist.

Exclusion Criteria:

* Those who have received systemic antibiotics within four weeks of starting the study.
* Those who have received systemic isotretinoin within six weeks of starting the study.
* Those with seborrheic dermatitis, rosacea, or polycystic ovary syndrome
* Those who are pregnant, prisoners or cognitively impaired.
* Those subjects who are currently using proton pump inhibits (as studies have shown this may impact the gut microbiome) (4)
* Those who have a BMI greater than >30 kg/m2, as studies have shown a reduction in the variability of intestinal microbes within this population (5).
* Those who have initiated or changed brand of oral contraceptive pill within 4 weeks of starting the study.
* Those who have autoimmune disorders as this group has been shown to have an altered microbiome (6)
* Those who have diabetes (6), immunodeficiencies (7), inflammatory bowel disease (6), hypercholesterolemia, as these groups have been shown to have altered gut microbiomes
* Those who have taken oral probiotic supplements (8) within 4 weeks of starting the study
* Given the nature of the instructions that need to be adhered to for accurate collection of samples and this data, non-English speaking individuals will be excluded from this pilot study.
* Allergies to the tetracycline group of antibiotics
* Those who do not fit the inclusion criteria

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in the diversity of the gut microbiome in those with and without acne. | 2 years
  The diversity will be evaluated by assessing the Bray-Curtis dissimilarity index and the Shannon diversity of the bacterial DNA in the gut microbiome.
Change in the diversity of the gut microbiome before and after the treatment of doxycycline in those with acne. | 2 years
  The diversity will be evaluated by assessing the Bray-Curtis dissimilarity index and the Shannon diversity of the bacterial DNA in the gut microbiome.

SECONDARY OUTCOMES:
Change in global acne grade score | 2 years
Change in the investigator global assessment of acne | 2 years
Change in the lesion count of inflammatory and non-inflammatory lesions | 2 years
Change in the diversity of the skin microbiome in those with and without acne | 2 years
  The diversity will be evaluated by assessing the Bray-Curtis dissimilarity index and the Shannon diversity of the bacterial DNA in the gut microbiome.
Change in the diversity of the skin microbiome before and after treatment with doxycycline in those with acne | 2 years
  The diversity will be evaluated by assessing the Bray-Curtis dissimilarity index and the Shannon diversity of the bacterial DNA in the gut microbiome.
Change in the diversity of the skin lipidome in those with and without acne | 2 years
  The lipid profile will include quantitation of the fatty acid profiles and presence of long chain fatty acids and short chain fatty acids.
Change in the skin lipidome before and after treatment with doxycycline in those with acne | 2 years
  The lipid profile will include quantitation of the fatty acid profiles and presence of long chain fatty acids and short chain fatty acids.
Change in the diversity of the blood lipidome in those with and without acne | 2 year
  The lipid profile will include quantitation of the fatty acid profiles and presence of long chain fatty acids and short chain fatty acids.
Change in the blood lipidome before and after treatment with doxycycline in those with | 2 years
  The lipid profile will include quantitation of the fatty acid profiles and presence of long chain fatty acids and short chain fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD MS CAT, Principal Investigator — UCDavis
Locations (1):
- UC Davis Dept of Dermatology, Sacramento, California, United States